CLINICAL TRIAL: NCT03285438
Title: REduced Dose Versus Full-dose of Direct Oral Anticoagulant After uNprOvoked Venous thromboEmbolism. The RENOVE Open-label, Randomized, Controlled Trial.
Brief Title: REduced Dose Versus Full-dose of Direct Oral Anticoagulant After uNprOvoked Venous thromboEmbolism.
Acronym: RENOVE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: University Hospital of Saint-Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 29BRC17.0125
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Venous Thromboembolism
Keywords: Venous Thromboembolism; Anticoagulant; Direct oral anticoagulant; risk of recurrent venous thromboembolism; anticoagulant-related bleeding
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Intervention Model Description: The trial is designed as an academic, multicenter, open, with blind evaluation (PROBE), randomized, parallel arm, controlled.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduced dose of DOAC (Experimental): A reduced dose of DOAC (apixaban 2.5 mg twice daily or rivaroxaban 10 mg once daily) during a mean follow-up period of 36 months (12 to 65 months)
  Interventions: Drug: Reduced dose of DOAC
- Full dose of DOAC (Active Comparator): A full dose of DOAC (Apixaban 5 mg twice daily or Rivaroxaban 20 mg once daily) during a mean follow-up period of 36 months (12 to 65 months).
  Interventions: Drug: Full dose of DOAC

INTERVENTIONS:
Drug: Reduced dose of DOAC — The patient will receive apixaban 2.5 mg twice daily or rivaroxaban 10 mg once daily during a mean follow-up period of 36 months (12 to 65 months)
  Arms: Reduced dose of DOAC
Drug: Full dose of DOAC — The patient will receive apixaban 5 mg twice daily or Rivaroxaban 20 mg once daily during a mean follow-up period of 36 months (12 to 65 months)
  Arms: Full dose of DOAC

SUMMARY:
Patients with unprovoked venous thromboembolism (VTE) or VTE associated with persistent risk factors have a high risk of recurrence after stopping anticoagulation. In these patients, international guidelines recommend indefinite anticoagulation. However, prolonged use of warfarin or DOAC at therapeutic dose is associated with a significant risk of bleeding. Consequently, it has been hypothesized that extended anticoagulation at lower dosage might be as effective as and safer than full dose of anticoagulation. However, low-dose warfarin (INR 1.5-2) was less effective and not safer than conventional dose warfarin (INR 2-3).

Low dose of DOAC has the potential to validate this hypothesis. In a first randomized trial comparing full-dose or low-dose apixaban with a placebo during an additional one year of anticoagulation in patients where physicians were uncertain for prolonging anticoagulation ("Amplify-extension trial"), low-dose apixaban was more effective than placebo without any major concern regarding safety and possibly as effective as and safer than full-dose apixaban; in a second randomized trial comparing full-dose or low-dose rivaroxaban with aspirin, during an additional one year of anticoagulation in patients where physicians were uncertain for prolonging anticoagulation ("Einstein-Choice trial"), low-dose rivaroxaban was more effective than aspirin without any major concern regarding safety and possibly as effective as and safer than full-dose rivaroxaban. However, these two studies were not designed and powered to demonstrate non-inferiority on efficacy and superiority on safety of a reduced dose of DOAC versus a full dose DOAC and the selected population did not have strong indications for indefinite anticoagulation. Thus, there is currently no evidence to recommend a reduced dose rather than a full dose of DOAC for extended therapy in patients at high risk of recurrent VTE. Consequently, a randomized trial comparing low-dose DOAC with full-dose DOAC therapy in patients at high risk of recurrent VTE is needed and justified.

Main hypothesis:

After VTE at high risk of recurrence initially treated during 6 (-15 days) to 24 (+ 3 months) uninterrupted months, a reduced dose of DOAC will be non-inferior to a full dose of DOAC in terms of recurrent VTE during extended anticoagulation phase.

DETAILED DESCRIPTION:
Patients with unprovoked venous thromboembolism (VTE) or VTE associated with persistent risk factors have a high risk of recurrence after stopping anticoagulation. In the "PADIS-PE" trial comparing an additional 18 months of warfarin (target international normalized ratio (INR) from 2 to 3) versus placebo in 371 patients who have completed 6 months of anticoagulation for a first unprovoked pulmonary embolism, the PADIS-PE trial confirmed that prolonged warfarin therapy was highly effective for preventing recurrent VTE but that benefit was lost after stopping anticoagulation. In another trial, similar findings had been reported using direct oral anticoagulants (DOAC) at therapeutic dose. These results reinforce international recommendation for indefinite anticoagulation in patients at high risk of recurrent VTE (unprovoked VTE, recurrent VTE or persistent risk factors).

However, prolonged use of warfarin or DOAC at therapeutic dose is associated with a significant risk of bleeding. Consequently, it has been hypothesized that extended anticoagulation at lower dosage might be as effective as and safer than full dose of anticoagulation. However, low-dose warfarin (INR 1.5-2) was less effective and not safer than conventional dose warfarin (INR 2-3).

Low dose of DOAC has the potential to validate this hypothesis. First, DOACs have been shown to be as effective as and safer than warfarin (INR 2-3) during the first 6 months of anticoagulation after an acute VTE. Second, in a first randomized trial comparing full-dose or low-dose apixaban with a placebo during an additional one year of anticoagulation in patients where physicians were uncertain for prolonging anticoagulation ("Amplify-extension trial"), low-dose apixaban was more effective than placebo without any major concern regarding safety and possibly as effective as and safer than full-dose apixaban; in a second randomized trial comparing full-dose or low-dose rivaroxaban with aspirin, during an additional one year of anticoagulation in patients where physicians were uncertain for prolonging anticoagulation ("Einstein-Choice trial"), low-dose rivaroxaban was more effective than aspirin without any major concern regarding safety and possibly as effective as and safer than full-dose rivaroxaban. However, these two studies were not designed and powered to demonstrate non-inferiority on efficacy and superiority on safety of a reduced dose of DOAC versus a full dose DOAC and the selected population did not have strong indications for indefinite anticoagulation. Thus, there is currently no evidence to recommend a reduced dose rather than a full dose of DOAC for extended therapy in patients at high risk of recurrent VTE. Consequently, a randomized trial comparing low-dose DOAC with full-dose DOAC therapy in patients at high risk of recurrent VTE is needed and justified.

Main hypothesis:

After VTE at high risk of recurrence initially treated during 6 (-15 days) to 24 (+3 months) uninterrupted months, a reduced dose of DOAC will be non-inferior to a full dose of DOAC in terms of recurrent VTE during extended anticoagulation phase.

Design

The "RENOVE" trial is designed as an academic, multicenter, open, with blind evaluation (PROBE), randomized, parallel arm, controlled, trial sponsored by the Brest University Hospital Center. Patients meeting the inclusion criteria will be randomized at visit 1 (day 0) and allocated to receive:

* either a reduced dose of DOAC (apixaban 2.5 mg twice daily or rivaroaxaban 10 mg once daily) during a mean follow-up period of 36 months.
* or a full dose of DOAC (Apixaban 5 mg twice daily or Rivaroxaban 20 mg once daily) during a mean follow-up period of 36 months.

The study is powered to demonstrate the following hypotheses using a three steps hierarchical analysis:

* Primary hypothesis: non-inferiority of a reduced dose of DOAC as compared to a full dose of DOAC on the risk of recurrent VTE;
* Secondary hypothesis: in case of the confirmation of the previous hypothesis, superiority of a reduced dose of DOAC on the risk of major or clinically relevant non-major bleeding.
* Third hypothesis: in case of the confirmation of the previous hypothesis, superiority of a reduced dose of DOAC on the risk of the composite of recurrent VTE, major bleeding or clinically relevant non major bleeding.

Randomization will be centralized and stratified on:

* Center
* Type of DOAC
* antiplatelet agent taking

At visit 1, patients will have a therapeutic education and they will be instructed to call research team in case of any medical event during the study treatment period. Follow-up visits will be planned at 3, 6, 12 months and every 6 months until study end (i.e.; after the last included patient has achieved 12-month of study treatment period).

All critical events will be adjudicated by an independent adjudication committee blinded from the treatment allocation. A data safety board will be constituted and will meet on a regular basis. Duration of each patient's participation will be on average 36 months (12 months for the last included patient) and a total duration of the study is expected for 65 months.

Objectives:

* Main Objective

  • To demonstrate that a reduced dose of DOAC is non-inferior to a full dose of DOAC for the risk of recurrent VTE during the during a mean study treatment period of 36 months in patients with VTE that warrants indefinite anticoagulation and who have been initially treated for 6 (-15 days) to 24 (+3 months) uninterrupted months.
* Secondary Objectives

  • Key secondary objectives: if the main objective is verified, key secondary objectives are to demonstrate the superiority of a reduced dose of DOAC over a full dose of DOAC during a mean study treatment period of 36 months :
* on the risk of major or CRNMB and, if confirmed,
* on the composite of recurrent VTE, major bleeding or CRNMB.

  • Other secondary objectives:
* To evaluate the benefit of a reduced dose of DOAC on the risk of major bleeding during a mean study treatment period of 36 months
* To evaluate the benefit of a reduced dose of DOAC on the composite outcome of recurrent VTE and major bleeding during a mean study treatment period of 36 months
* To determine the impact of a reduced dose of DOAC on deaths of all causes and deaths related to recurrent VTE or major bleeding during a mean study treatment period of 36 months
* To evaluate dyspnea and post-thrombotic syndrome (villalta score)(65).
* To evaluate compliance treatment using the Girerd auto-questionnaire
* To analyse the treatment effect on recurrent VTE and major bleeding and CRNM among predefined sub-groups (screening for heterogeneity among predefined strata).

Sample size justification

A- Initial hypothesis before starting enrolment in the RENOVE study:

The study is powered to demonstrate the following hypotheses using a three steps hierarchical analysis:

* Primary hypothesis: non-inferiority of a reduced dose of DOAC as compared to a full dose of DOAC on the risk of recurrent VTE. Based on an expected rate of recurrent VTE of 2%/year (4% during the entire study period) in each group and a requirement that the study would have 90% power to exclude a hazard ratio of 1.7 for the primary outcome with a reduced dose of DOAC, at a two-sided alpha level of 0.05, 1030 patients need to be included in each treatment group.
* Secondary hypothesis: in case of the confirmation of the previous hypothesis, superiority of a reduced dose of DOAC on the risk of major or clinically relevant non-major bleeding. Assuming an estimated incidence in the warfarin group of 10% in the entire study period and a reduction in the relative risk of at least 35% with a reduced dose of DOAC as compared with a full dose of DOAC, 966 patients in each group for the study to have 80% power to show the superiority of a reduced dose of DOAC over a full dose of DOAC, at a two-sided alpha level of 0.05.
* Third hypothesis: in case of the confirmation of the previous hypothesis, superiority of a reduced dose of DOAC on the risk of the composite of recurrent VTE, major bleeding or clinically relevant non major bleeding. Assuming an estimated incidence in the full dose DOAC group of 14% and 10% in the a reduced dose of DOAC group in the entire study period, 1029 patients in each group for the study to have 80% power to show the superiority of a reduced dose of DOAC over a full dose of DOAC, at a two-sided alpha level of 0.05.

Taking in account 5% of loss to follow-up, a total of 2200 patients are required in order to be able to confirm these three conditional hypotheses.

All estimates were calculated based on major randomized trials on extended anticoagulation in VTE patients.

B- New hypothesis based on observed primary endpoint at 2147 included patients:

On February, 12th 2021, 27 recurrent VTE, all adjudicated, occurred on 2147 included patients, during a mean follow-up of 12 months.

* From 0 to 12 months, there were 15 recurrent VTE in 2147 patients during this period (0.7%); and
* from 12 to 24 months, there were 12 recurrent VTE in 1551 patients during this period (0.8%).
* The incidence of recurrence seems to be linear, with 0.75% patients with recurrent VTE during a mean follow-up of 12 months. Consequently, the expected proportion of recurrent VTE during 24 months will be 1.5% and not 4% as previously expected before study started.
* The scientific committee, blinded of treatment group, decided to increase both the number of sample size and the follow-up with a new "first" hypothesis on recurrent VTE:
* New First hypothesis: same non inferiority of a reduced dose of DOAC compared to a full dose of DOAC on the risk of recurrent VTE. Based on a new expected rate of recurrent VTE of 3% in each group during the entire study period for the same power (90%) and the same alpha level (two-side alpha level of 0.05), with a similar hazard ratio non-inferiority margin, i.e., 1.7, 1387 patients need to be included in each treatment group. Thus, a total of 2774 patients need to be recruited, which correspond to 574 patients in addition to 2200. Keeping in mind that the recruitment is 60 patients per months, the time to recruit 574 additional patients will take 6 months. We will stop the study after the last included patient has been followed at least 12 months. Thus, the study is prolonged by 18 additional months (6 to 8 months recruitment + 12-month follow up of the last patient).

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years
* Patients with indications for long-term anticoagulation after VTE (i.e.; symptomatic PE or proximal DVT) initially treated during 6 (-15 days) to 24 months (+ 3 months) :

  * Patients with multiple episodes of VTE, or
  * Patients with a first episode of unprovoked* VTE
  * Patients with VTE associated with persistent risk factor**, or
  * Patients for whom clinicians feel that indefinite anticoagulation is warranted
* Social security affiliation.

Exclusion Criteria:

* Known allergy to rivaroxaban and apixaban, allergy to any of the excipients
* Indication for therapeutic dose anticoagulant therapy
* Unable or refusal to give informed consent
* Isolated distal DVT
* HERDOO2 score ≤ 1
* Indication for anticoagulation other than DVT or PE (e.g.; atrial fibrillation, mechanic valves…)
* Treatment with investigational drug in the past 1 month except for patients benefiting from an anticoagulant at therapeutic doses for the initial pathology
* Interruption of anticoagulation for 14 days or more before the inclusion
* Chronic liver disease or chronic hepatitis
* Patient considered at high risk of bleeding (eg: previous gastro-intestinal tract bleeding in the past three months, uncontrolled hypertension, etc.)
* Renal insufficiency with creatinine <25 ml / min on Cockcroft and Gault formula
* Antiphospholipid syndrome
* Dual anti-platelet therapy or aspirin at dosage >100 mg per day
* Concomitant use of a strong inhibitor of cytochrome P-450 3A4 (CYP3A4) (e.g., a protease inhibitor for human immunodeficiency virus infection or azole-antimycotics agents ketoconazole, itraconazole, voriconazole, posaconazole) or a CYP3A4 inducer (e.g., rifampin, carbamazepine, or phenytoin),
* Active cancer of less than 6 months
* Active pregnancy or expected pregnancy
* No effective contraception in women of childbearing age
* Life expectancy <12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2774 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
Recurrent VTE | during a mean study treatment period of 36 months
  Adjudicated symptomatic objectively confirmed recurrent VTE (non fatal or fatal VTE) during the study treatment period.

SECONDARY OUTCOMES:
Major and clinically relevant non major bleeding | during a mean study treatment period of 36 months
  Adjudicated major bleeding (as defined by the criteria of the International Society of Thrombosis and Haemostasis) or clinically relevant non major bleeding during the study treatment period
The composite of recurrent VTE or major bleeding or non major clinically relevant bleeding | during a mean study treatment period of 36 months
  The composite of adjudicated recurrent VTE or major bleeding or non major clinically relevant bleeding during the study treatment period will be adjudicated
Mortality | during a mean study treatment period of 36 months
  Mortality of other cause than recurrent VTE or major or clinically relevant non major bleeding during the study treatment period will be adjudicated
Compliance | during a mean study treatment period of 36 months
  Treatment compliance will be evaluated
Treatment effect | during a mean study treatment period of 36 months
  The heterogeneity of the treatment effect on predefined strata will be evaluated
Arterial cardio-vascular events | during a mean study treatment period of 36 months
  The arterial cardio-vascular events (myocardial infarction, stroke, cardio-vascular complication other than VTE) will be evaluated

CONTACTS AND LOCATIONS:
Locations (38):
- France (38):
  - CHU Amiens-Picardie, Amiens
  - CHU Angers, Angers
  - CH d'Arras, Arras
  - CHU de Besançon - Hôpital Jean Minjoz, Besançon
  - CH Bordeaux, Bordeaux
  - HIA Brest, Brest
  - CHRU de Brest, Brest
  - Clinique de Clapiers, Castelnau-le-Lez
  - HIA Percy, Clamart
  - Cabinet médical, Clapiers
  - CHU de Clermont Ferrand - Hôpital Gabriel Montpied, Clermont-Ferrand
  - APHP Hôpital Louis Mourier, Colombes
  - CHU de Dijon, Dijon
  - CHU de Grenoble - Hôpital Nord Michallon, Grenoble
  - GH Le Havre, Le Havre
  - CH Le Mans, Le Mans
  - CHU de Limoges - Hôpital de Dupuytren, Limoges
  - CH Morlaix, Morlaix
  - Chru Nancy, Nancy
  - CHU de Nantes, Nantes
  - CHU de Nice - Hôpital Pasteur, Nice
  - CHU Nîmes, Nîmes
  - CHR Orléans, Orléans
  - Hôpital de Cochin, Paris
  - HEGP, Paris
  - CHU Paris Nord Val de Seine, Paris
  - Kremlin Bicêtre, Paris
  - CH de Périgueux, Périgueux
  - CH de Quimper, Quimper
  - CHU de Rennes - Hôpital Sud, Rennes
  - CHU de ROUEN, Rouen
  - CH de Saint Brieuc - Hôpital Yves Le Foll, Saint-Brieuc
  - CHU de Saint Etienne - Hôpital Nord, Saint-Etienne
  - CH de Toulon - Hôpital Sainte-Musse, Toulon
  - HIA Sainte-Anne, Toulon
  - CHU de Toulouse - Hôpital de Rangueil, Toulouse
  - CHU de Tours - Hôpital Trousseau, Tours
  - CH Valenciennes, Valenciennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Couturaud F, Schmidt J, Sanchez O, Ballerie A, Sevestre MA, Meneveau N, Bertoletti L, Connault J, Benhamou Y, Constans J, Quemeneur T, Lapebie FX, Pernod G, Picart G, Elias A, Doutrelon C, Neveux C, Khider L, Roy PM, Zuily S, Falvo N, Lacroix P, Emmerich J, Mahe I, Boileau J, Yaici A, Le Jeune S, Stephan D, Plissonneau-Duquene P, Ray V, des Deserts MD, Belhadj-Chaidi R, Lamia B, Gruel Y, Presles E, Girard P, Tromeur C, Moustafa F, Rothstein V, Lacut K, Melac S, Barillot S, Mismetti P, Laporte S, Mottier D, Meyer G, Leroyer C; RENOVE Investigators. Extended treatment of venous thromboembolism with reduced-dose versus full-dose direct oral anticoagulants in patients at high risk of recurrence: a non-inferiority, multicentre, randomised, open-label, blinded endpoint trial. Lancet. 2025 Mar 1;405(10480):725-735. doi: 10.1016/S0140-6736(24)02842-3. PMID 40023651